CLINICAL TRIAL: NCT05009251
Title: Using Explainable AI Risk Predictions to Nudge Influenza Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Geisinger Clinic (Other); Massachusetts Institute of Technology (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0483; P30AG034532 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Influenza; Vaccination; Health Promotion; Health Behavior; Risk Reduction
Keywords: Flu Vaccine; Choice Architecture; Machine Learning; Perceived Credibility; Personalized Risk Factors; Flu Complications
MeSH Terms: conditions — Influenza, Human; Health Behavior; Risk Reduction Behavior | interventions — Numbers Needed To Treat

STUDY DESIGN:
Intervention Model Description: Patients from the high-risk sample will be randomly assigned to one of five arms:
  * No-Contact Control Arm
  * Reminder Control Arm
  * High Risk Only Arm
  * High Risk with Explanation Based on Medical Records Arm
  * High Risk with Explanation Based on Algorithm Arm
Who Masked: Care Provider
Masking Description: Providers who prescribe vaccination and diagnose conditions will not be randomized to study arms or informed of patient assignment. Although patients will not be explicitly informed which arm they have been randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No-Contact Control (No Intervention): Subjects in the no-contact control arm will receive no additional pro-vaccination intervention beyond the health system's normal efforts. Although some patients are currently targeted for flu vaccination encouragement due to a conventional non-ML assessment that they are at high risk for complications, these patients are not told that they are at high risk or that they have been targeted.
- Reminder Control (Experimental): Subjects in the reminder control arm will receive messages reminding them to get the flu shot without being advised of their risk status.
  Interventions: Behavioral: Reminder
- High Risk Only (Experimental): Subjects in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications, without specifying how or why the health system believes this to be the case.
  Interventions: Behavioral: Reminder; Behavioral: Risk reduction
- High Risk with Explanation Based on Medical Records (Experimental): Subjects in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications via review of their medical records and will be provided a human-understandable short list of the top factors from their medical record that explain their risk.
  Interventions: Behavioral: Reminder; Behavioral: Risk reduction; Behavioral: Medical records-based recommendation
- High Risk with Explanation Based on Algorithm (Experimental): Subjects in this treatment arm will receive messages telling them they have been identified to be at high risk for flu complications via analysis of their medical records by a computer algorithm and will be provided a human-understandable short list of the top factors from their medical record that explain their risk.
  Interventions: Behavioral: Reminder; Behavioral: Risk reduction; Behavioral: Medical records-based recommendation; Behavioral: Algorithm-based recommendation

INTERVENTIONS:
Behavioral: Reminder — Mailed letter, short message service (SMS) text, and/or patient portal message
  Arms: High Risk Only; High Risk with Explanation Based on Algorithm; High Risk with Explanation Based on Medical Records; Reminder Control
Behavioral: Risk reduction — Mailed letter, SMS, and/or patient portal message
  Arms: High Risk Only; High Risk with Explanation Based on Algorithm; High Risk with Explanation Based on Medical Records
Behavioral: Medical records-based recommendation — Mailed letter, SMS, and/or patient portal message
  Other Names: Credibility
  Arms: High Risk with Explanation Based on Algorithm; High Risk with Explanation Based on Medical Records
Behavioral: Algorithm-based recommendation — Mailed letter, SMS, and/or patient portal message
  Other Names: Credibility
  Arms: High Risk with Explanation Based on Algorithm

SUMMARY:
The study team previously demonstrated that patients are more likely to receive flu vaccine after learning that they are at high risk for flu complications. Building on this past work, the present study will explore whether providing reasons that patients are considered high risk for flu complications (a) further increases the likelihood they will receive flu vaccine and (b) decreases the likelihood that they receive diagnoses of flu and/or flu-like symptoms in the ensuing flu season. It will also examine whether informing patients that their high-risk status was determined by analyzing their medical records or by an artificial intelligence (AI) / machine-learning (ML) algorithm analyzing their medical records will affect the likelihood of receiving the flu vaccine or diagnoses of flu and/or flu-like symptoms.

DETAILED DESCRIPTION:
Geisinger has partnered with Medial EarlySign and developed an ML algorithm to identify patients at risk for serious (moderate to severe) flu-associated complications on the basis of their existing electronic health record (EHR) data. Geisinger will apply this algorithm to current patients during the 2021-22 flu season.

This study will evaluate the effect of contacting patients identified as high risk with special messages to encourage vaccination. These communications will inform patients they are at high risk with either (a) no additional explanation, (b) an explanation that this determination comes from an analysis of their medical records, along with a short list of the top factors from their medical record that explain their risk, and (c) the additional explanation that an AI or ML algorithm made this determination, along with a short list of the top factors from their medical record that explain their risk.

Included in the study will be current Geisinger patients 18+ years of age with no contraindications for flu vaccine and who have been assessed by the Medial algorithm and assigned a risk score. The primary study outcomes will be the rates of flu vaccination and flu diagnosis during the 2020-21 season by targeted patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Current Geisinger patient at the time of study
* Falls in the top 10% of patients at highest risk, as identified by the flu-complication risk scores of machine learning algorithm (which operates on coded EHR data)

Exclusion Criteria:

* Has contraindications for flu vaccination
* Has opted out of receiving communications from Geisinger via all of the modalities being tested

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45061 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Meyer, PhD JD, Principal Investigator — Geisinger Clinic; Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data and code are available in the below repository in the folder ClinicalTrials.gov data/Study 2.
URL: https://osf.io/mqbux/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Started | 9017 | 9013 | 9011 | 9003 | 9017
Completed | 8892 | 8886 | 8868 | 8864 | 8883
Not Completed | 125 | 127 | 143 | 139 | 134
Not completed — Protocol Violation | 100 | 105 | 119 | 120 | 119
Not completed — Death | 25 | 22 | 24 | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm | Total
Number analyzed (Participants) | 9017 | 9013 | 9011 | 9003 | 9017 | 45061
Age, Customized [Count of Participants; unit: Participants]
  >=18 years and <65 | 6018 | 5984 | 6049 | 6001 | 6004 | 30056
  >=65 | 2999 | 3029 | 2962 | 3002 | 3013 | 15005
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6038 | 6121 | 6107 | 6086 | 6140 | 30492
  Male | 2979 | 2892 | 2904 | 2917 | 2877 | 14569
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 381 | 351 | 374 | 353 | 365 | 1824
  Not Hispanic or Latino | 8608 | 8635 | 8607 | 8627 | 8630 | 43107
  Unknown or Not Reported | 28 | 27 | 30 | 23 | 22 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 19 | 14 | 16 | 16 | 76
  Asian | 27 | 21 | 23 | 26 | 27 | 124
  Native Hawaiian or Other Pacific Islander | 15 | 12 | 12 | 16 | 20 | 75
  Black or African American | 348 | 286 | 300 | 330 | 300 | 1564
  White | 8596 | 8660 | 8648 | 8602 | 8636 | 43142
  Unknown or Not Reported | 20 | 15 | 14 | 13 | 18 | 80

OUTCOME MEASURES:

1. Primary Outcome: Flu Vaccination at 2 Weeks After Final Outreach Date
Description: Received flu vaccination
Time Frame: Within 2 weeks of the final outreach date, 57 days (8.14 weeks) after the study start
Population: Patients were excluded from analyses if they died before or during the study, if they were contraindicated for flu vaccine, if they were sent protective risk reasons, or if they were vaccinated prior to the study beginning. See the Statistical Analysis Plan for more information on exclusions.
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  Not Vaccinated | 5798 | 5715 | 5560 | 5583 | 5662
  Vaccinated | 2668 | 2807 | 2938 | 2887 | 2863
Statistical Analysis 1: Comparison: Reminder Control vs High Risk Only vs High Risk With Explanation Based on Medical Records vs High Risk With Explanation Based on Algorithm; This analysis compared groups that were informed they were high risk (High Risk Only, High Risk Based on Medical Records, High Risk Based on Algorithm) to Reminder Control patients who were sent messages that did not disclose their risk status. Null hypothesis: messages that inform patients they are high risk do not increase flu vaccination rate vs. messages that do not disclose risk status; Alternative hypothesis: messages that inform patients they are high risk increase flu vaccination rate; Test type: Superiority; p = .054, Regression, Linear
Statistical Analysis 2: Comparison: No-Contact Control vs High Risk Only vs High Risk With Explanation Based on Medical Records vs High Risk With Explanation Based on Algorithm; This analysis compared groups that were informed they were high risk (High Risk Only, High Risk Based on Medical Records, High Risk Based on Algorithm) to No-Contact Control patients who were not sent messages. Null hypothesis: messages that inform patients they are high risk do not increase flu vaccination rate relative to no messages; Alternative hypothesis: messages that inform patients they are high risk increase flu vaccination rate; Test type: Superiority; p < .001, Regression, Linear
Statistical Analysis 3: Comparison: High Risk Only vs High Risk With Explanation Based on Medical Records vs High Risk With Explanation Based on Algorithm; This analysis compared groups who received messages including risk reasons (High Risk Based on Medical Records, High Risk Based on Algorithm) to messages that mentioned patients' risk status but do not include reasons (High Risk Only). Null hypothesis: messages that include risk reasons do not increase flu vaccination rate relative to high-risk messages that do not include risk reasons; Alternative hypothesis: messages including risk reasons are more effective at increasing vaccination rates; Test type: Superiority; p = .240, Regression, Linear
Statistical Analysis 4: Comparison: No-Contact Control vs Reminder Control; Null hypothesis: flu-shot messages that do not mention high-risk status do not increase vaccination relative to no messages; Alternative hypothesis: flu shot messages that do not mention high-risk status increase flu shots relative to no messages; Test type: Superiority; p = .047, Regression, Linear
Statistical Analysis 5: Comparison: High Risk Only vs High Risk With Explanation Based on Medical Records; Null hypothesis: High Risk Only and High Risk Based on Medical Records messages are equally effective at promoting flu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High Risk Only and High Risk Based on Medical Records; Test type: Superiority; p = .781, Regression, Linear — Pairwise comparisons between high-risk messages (Analyses 5, 6 and 7) were analyzed in the same regression. Reported p-values were adjusted using Tukey's HSD test
Statistical Analysis 6: Comparison: High Risk Only vs High Risk With Explanation Based on Algorithm; Null hypothesis: High Risk Only and High Risk Based on Algorithm messages are equally effective at promoting flu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High Risk Only and High Risk Based on Algorithm; Test type: Superiority; p = .361, Regression, Linear — [p-value comment as in outcome 1, analysis 5]
Statistical Analysis 7: Comparison: High Risk With Explanation Based on Medical Records vs High Risk With Explanation Based on Algorithm; Null hypothesis: High Risk Based on Medical Records and High Risk Based on Algorithm messages are equally effective at promoting flu vaccinations; Alternative hypothesis: there is a difference in effectiveness between High Risk Based on Medical Records and High Risk Based on Algorithm; Test type: Superiority; p = .770, Regression, Linear — [p-value comment as in outcome 1, analysis 5]

2. Secondary Outcome: Flu Vaccination at 9 Weeks After Final Outreach Date
Description: Received a flu vaccination
Time Frame: Within 9 weeks of the final outreach date, 106 days (15.14 weeks) after the study start
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  Not Vaccinated | 5180 | 5093 | 4973 | 4935 | 5076
  Vaccinated | 3286 | 3429 | 3525 | 3535 | 3449

3. Secondary Outcome: Flu Diagnosis
Description: Received a "high confidence flu" diagnosis (with positive polymerase chain reaction [PCR]/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test)
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Time Frame: 8 months (between September 9, 2021 and April 30, 2022)
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  No flu diagnosis | 8336 | 8382 | 8365 | 8346 | 8385
  Flu diagnosis | 130 | 140 | 133 | 124 | 140

4. Secondary Outcome: Flu Complications
Description: Diagnosed with flu-related complications
Time Frame: 11 months (between September 9, 2021 and July 31, 2022)
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  No flu complications | 5916 | 5904 | 5910 | 5861 | 5853
  Flu complications | 2550 | 2618 | 2588 | 2609 | 2672

5. Secondary Outcome: Healthcare Utilization
Description: Visited ER or was hospitalized
  NOTE: Our prespecified outcome was description was "Visited ER, was hospitalized, or had flu-related insurance claims." We did not receive claims data, so this outcomes includes only ER visits and hospitalizations.
Time Frame: 11 months (between September 9, 2021 and July 31, 2022)
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  No utilization | 5203 | 5221 | 5205 | 5160 | 5311
  Utilization | 3263 | 3301 | 3293 | 3310 | 3214

6. Other Pre Specified Outcome: Flu Vaccination at 2 Weeks After Final Outreach Date by Gender
Description: Received a flu vaccination
Time Frame: Within 2 weeks of the final outreach date, 57 days (8.14 weeks) after the study start
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  Female: number analyzed (Participants) | 5670 | 5794 | 5746 | 5740 | 5816
  Female | 1740 | 1840 | 1933 | 1878 | 1933
  Male: number analyzed (Participants) | 2796 | 2728 | 2752 | 2730 | 2709
  Male | 928 | 967 | 1005 | 1009 | 930

7. Other Pre Specified Outcome: Flu Vaccination at 2 Weeks After Final Outreach Date by Race
Description: Received Flu Vaccination
Time Frame: Within 2 weeks of the final outreach date, 57 days (8.14 weeks) after the study start
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 11 | 16 | 10 | 16 | 15
  American Indian or Alaska Native | 2 | 3 | 1 | 2 | 7
  Asian: number analyzed (Participants) | 26 | 18 | 22 | 24 | 26
  Asian | 8 | 5 | 7 | 12 | 7
  Black: number analyzed (Participants) | 337 | 277 | 284 | 316 | 290
  Black | 67 | 51 | 68 | 61 | 49
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 14 | 12 | 10 | 15 | 17
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 1 | 6 | 3
  Unknown: number analyzed (Participants) | 20 | 14 | 14 | 13 | 14
  Unknown | 1 | 5 | 4 | 5 | 1
  White: number analyzed (Participants) | 8058 | 8185 | 8158 | 8086 | 8163
  White | 2586 | 2742 | 2857 | 2801 | 2796

8. Other Pre Specified Outcome: Flu Vaccination at 2 Weeks After Final Outreach Date by Ethnicity
Description: Received flu vaccination
Time Frame: Within 2 weeks of the final outreach date, 57 days (8.14 weeks) after the study start
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
Number analyzed (Participants) | 8466 | 8522 | 8498 | 8470 | 8525
Participants
  Hispanic or Latino: number analyzed (Participants) | 362 | 335 | 355 | 336 | 347
  Hispanic or Latino | 76 | 76 | 68 | 78 | 71
  Not Hispanic or Latino: number analyzed (Participants) | 8076 | 8160 | 8116 | 8113 | 8156
  Not Hispanic or Latino | 2578 | 2722 | 2865 | 2804 | 2784
  Unable to Obtain: number analyzed (Participants) | 28 | 27 | 27 | 21 | 22
  Unable to Obtain | 14 | 9 | 5 | 5 | 8

ADVERSE EVENTS:
Time Frame: Roughly 1 month (9/9/21 - 10/7/21)
Description: This is a minimal risk study, and has received expedited IRB review in keeping with 45 CFR § 46.110. EHR and claims data will report inputs (i.e., the subject's assigned arm) and outcomes (i.e., flu vaccination, flu diagnosis, flu-like symptoms). We therefore did not monitor the data for AE/SAEs. However, on 10/7/2021, we completed a data pull with an updated death record check, and patients who died during the study as of that data pull are indicated under All-Cause Mortality.
Arm/Group | No-Contact Control | Reminder Control | High Risk Only | High Risk With Explanation Based on Medical Records | High Risk With Explanation Based on Algorithm
All-Cause Mortality (participants affected / at risk) | 25/9017 | 22/9013 | 24/9011 | 19/9003 | 17/9017
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05009251/Prot_001.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT05009251/SAP_000.pdf